CLINICAL TRIAL: NCT03384966
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled Study to Assess the Pharmacodynamics, Pharmacokinetics, Tolerability, and Safety of a Single Subcutaneous Injection of ACT-246475 in Adults With Stable Coronary Artery Disease
Brief Title: A Medical Research Study to Evaluate the Effects of ACT-246475 in Adults With Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-076A201; 2017-003332-36 (EudraCT Number)
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2022-11

CONDITIONS: Stable Coronary Artery Disease
Keywords: Chronic coronary syndrome
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinding will apply to treatment (ACT-246475 vs placebo). The dose (8 mg vs 16 mg) will be single blinded (subject blinded). The site for the sub-cutaneous injection (thigh vs abdomen) will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Selatogrel 8 mg (Experimental): Selatogrel (ACT-246475) is given as a single subcutaneous dose of 8 mg administered in a volume of 0.8 mL. Administration will be performed at the investigational site by qualified personnel.
  Interventions: Drug: Selatogrel
- Selatogrel 16 mg (Experimental): Selatogrel (ACT-246475) is given as a single subcutaneous dose of 16 mg administered in a volume of 0.8 mL. Administration will be performed at the investigational site by qualified personnel.
  Interventions: Drug: Selatogrel
- Placebo (Placebo Comparator): Placebo matching ACT-246475 is supplied in sealed glass vials for reconstitution with water for injection. Placebo will be given as a single subcutaneous dose matching selatogrel to be administered in a volume of 0.8 mL. Administration will performed at the investigational site by qualified personnel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selatogrel — Selatogrel is a reversible P2Y12 receptor antagonist for subcutaneous administration. It is supplied in sealed glass vials at a strength of 20 mg. The vials with ACT-246475A (hydrochloride salt of ACT-246475) or matching placebo will be reconstituted with 1 mL of water for injection. Further dilution with 1 mL sodium chloride (NaCl) 0.9% will be performed for preparation of the dose of 8 mg selatogrel.
  Other Names: ACT-246475
  Arms: Selatogrel 8 mg
Drug: Placebo — Matching placebo for subcutaneous administration.
  Arms: Placebo
Drug: Selatogrel — Selatogrel is a reversible P2Y12 receptor antagonist for subcutaneous administration. It is supplied in sealed glass vials at a strength of 20 mg. The vials with ACT-246475A (hydrochloride salt of ACT-246475) will be reconstituted with 1 mL of water for injection.
  Other Names: ACT-246575
  Arms: Selatogrel 16 mg

SUMMARY:
The goal of this study is to find out if a drug called selatogrel (ACT-246475) can prevent platelets from binding together when administered by an injection under the skin in the thigh or in the belly. Another goal is to know how fast and for how long selatogrel (ACT-246475) works and if there is a difference if the drug is injected in the thigh or in the belly. This study will also help to find out more about the safety of this new drug.

DETAILED DESCRIPTION:
To investigate the pharmacodynamic (PD) and pharmacokinetic (PK) properties of selatogrel in patients with atherosclerotic disease, the present study will be conducted in patients with chronic coronary syndromes (CCS). Assessment in a population of patients with CCS allows better control and stability of concomitant treatments, and therefore more accurate characterization of the pharmacodynamic and pharmacokinetic profiles of selatogrel in the presence of background antiplatelet therapies.

The study will have 3 periods: a screening period of up to 21 days prior to randomization, a treatment period of 2 days from randomization (Day 1) to 24 hours post dose (Day 2), and a follow-up period from Day 3 to the safety follow-up telephone call 28 to 35 days after single administration of study drug (End-of-Study).

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Male and female subjects aged from 18-85 years, inclusive.
3. For women of childbearing potential: Negative urine pregnancy test at Visit 1 and at Visit 2 before randomization.
4. Stable Coronary artery disease (CAD) defined by the presence of any of the following conditions:

   1. History of CAD with coronary artery stenosis on coronary angiogram ≥50%.
   2. Previously documented myocardial infarction occurring more than 3 months prior to randomization.
5. Antiplatelet background therapy stable for at least 1 month prior to randomization.
6. Body weight ≥ 40.0 kg (88.2 lbs).

Main Exclusion Criteria:

1. Acute coronary syndrome, percutaneous coronary intervention or any intervention for peripheral artery disease within 3 months prior to randomization.
2. Acute ischemic stroke or transient ischemic attack (TIA) within 3 months prior to randomization.
3. Active internal bleeding, or medical history of recent (< 1 month) bleeding disorders or conditions associated with high risk of bleeding (e.g., clotting disturbances, gastrointestinal bleed, hemoptysis).
4. Hemoglobin ≤ 10 g/dL at screening.
5. Loss of at least 250 mL of blood within 3 months of screening.
6. Use of anticoagulants (oral, parenteral) or fibrinolytic therapy within 24 h prior to screening (Visit 1).
7. Known platelet disorders (e.g., thrombasthenia, thrombocytopenia, von Willebrand disease).
8. Pregnant or breastfeeding women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (20):
- United States (7):
  - University of Florida (UF) Jacksonville, Jacksonville, Florida
  - Florida Hospital Tampa - Pepin Heart Institute, Tampa, Florida
  - NorthShore University, Chicago, Illinois
  - Indiana University School of Medicine - Krannert Institute of Cardiology, Indianapolis, Indiana
  - Inova Cardiology, Lutherville, Maryland
  - Mount Sinai Hospital (New York), New York, New York
  - Inova Center for Thrombosis Research and Translational Medicine, Falls Church, Virginia
- Institut de Cardiologie de Montréal, Montreal, Quebec, Canada
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- Universitats-Herzzentrum, Bad Krozingen, Germany
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Maastricht UMC, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
- National Heart Centre Singapore, Singapore, Singapore
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Uppsala University Hospital, Uppsala
- United Kingdom (3):
  - Freeman Hospital - Cardiothoracic Department, Newcastle upon Tyne
  - Sheffield Teaching Hospitals, Sheffield
  - East & North Hertfordshire NHS Trust - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Storey RF, Gurbel PA, Ten Berg J, Bernaud C, Dangas GD, Frenoux JM, Gorog DA, Hmissi A, Kunadian V, James SK, Tanguay JF, Tran H, Trenk D, Ufer M, Van der Harst P, Van't Hof AWJ, Angiolillo DJ. Pharmacodynamics, pharmacokinetics, and safety of single-dose subcutaneous administration of selatogrel, a novel P2Y12 receptor antagonist, in patients with chronic coronary syndromes. Eur Heart J. 2020 Sep 1;41(33):3132-3140. doi: 10.1093/eurheartj/ehz807. PMID 31994703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 24 Jan and 18 Sep 2018. Twenty sites in 8 countries screened 362 participants and 17 sites randomized 346 participants.
Pre-assignment Details: Of the 16 participants not randomized: 9 were ineligible; 4 withdrew consent; 1 was lost to follow-up, 1 was not randomized based on the physician's decision and 1 didn't complete screening within the protocol-defined window.
Groups:
- Selatogrel 8 mg: The study had 3 consecutive periods: the screening period, a treatment period and the follow-up period.
  A participant that met all inclusion criteria and none of the exclusion criteria was randomized.
  In the treatment period 8 mg of selatogrel (ACT-246475) was administered via a single subcutaneous injection either in the abdomen or the thigh.
  The follow-up period started on Day 3 and ended with the safety follow-up telephone call or visit (Day 35).
- Selatogrel 16 mg: The study had 3 consecutive periods: the screening period, a treatment period and the follow-up period.
  A participant that met all inclusion criteria and none of the exclusion criteria was randomized.
  In the treatment period 16 mg of selatogrel (ACT-246475) was administered via a single subcutaneous injection either in the abdomen or the thigh.
  The follow-up period started on Day 3 and ended with the safety follow-up telephone call or visit (Day 35).
- Placebo: The study had 3 consecutive periods: the screening period, a treatment period and the follow-up period.
  A participant that met all inclusion criteria and none of the exclusion criteria was randomized.
  In the treatment period placebo matching selatogrel was administered via a single subcutaneous injection either in the abdomen or the thigh.
  The follow-up period started on Day 3 and ended with the safety follow-up telephone call or visit (Day 35).
Period: Randomized at End of Screening Period
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Started | 115 | 115 | 116
Completed | 114 | 115 | 116
Not Completed | 1 | 0 | 0
Not completed — Physician decision due to adverse event | 1 | 0 | 0
Period: Treatment Period
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Started | 114 | 115 | 116
Thigh Administration | 57 | 57 | 58
Abdomen Administration | 57 | 58 | 58
Per-protocol Analysis Set (The per-protocol set includes all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).) | 96 | 90 | 93
Safety Analysis Set (The safety analysis set (SAF) includes all participants who received at least one dose of study treatment. Participants were evaluated according to the actual treatment they received.) | 114 | 115 | 116
Pharmacokinetic Analysis Set (The PK analysis set includes all participants from the SAF who have at least one plasma concentration measurement after administration of study treatment. Participants in the PK set were evaluated according to the actual treatment they received.) | 111 | 115 | 0
Completed | 114 | 115 | 116
Not Completed | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Started | 114 | 115 | 116
Completed | 113 | 115 | 116
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set - all participants that were randomized and who had study treatment administered.
Groups:
- Selatogrel 8 mg: Selatogrel (ACT-246475) 8 mg was administered as a single subcutaneous dose.
- Selatogrel 16 mg: Selatogrel (ACT-246475) 16 mg was administered as a single subcutaneous dose.
- Placebo: Matching placebo was administered as a single subcutaneous dose.
- Total: Total of all reporting groups
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo | Total
Number analyzed (Participants) | 114 | 115 | 116 | 345
Age, Categorical [Count of Participants; unit: Participants] — Population: Per-protocol set - all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full analysis set: <=18 years | 0 | 0 | 0 | 0
    Full analysis set: Between 18 and 65 years | 48 | 48 | 55 | 151
    Full analysis set: >=65 years | 66 | 67 | 61 | 194
    Per-protocol analysis set: number analyzed (Participants) | 96 | 90 | 93 | 279
    Per-protocol analysis set: <=18 years | 0 | 0 | 0 | 0
    Per-protocol analysis set: Between 18 and 65 years | 41 | 36 | 43 | 120
    Per-protocol analysis set: >=65 years | 55 | 54 | 50 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per-protocol set - all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  years
    Full analysis set | 64.8 (9.4) | 65.2 (8.5) | 64.9 (9.1) | 65.0 (9.0)
    Per-protocol analysis set: number analyzed (Participants) | 96 | 90 | 93 | 279
    Per-protocol analysis set | 64.4 (9.7) | 65.3 (8.8) | 65.1 (9.2) | 64.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Per-protocol set - all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full analysis set: Female | 20 | 26 | 23 | 69
    Full analysis set: Male | 94 | 89 | 93 | 276
    Per-protocol analysis set: number analyzed (Participants) | 96 | 90 | 93 | 279
    Per-protocol analysis set: Female | 16 | 17 | 16 | 49
    Per-protocol analysis set: Male | 80 | 73 | 77 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per-protocol set - all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full analysis set: Hispanic or Latino | 1 | 1 | 0 | 2
    Full analysis set: Not Hispanic or Latino | 113 | 114 | 116 | 343
    Full analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0
    Per-protocol analysis set: number analyzed (Participants) | 96 | 90 | 93 | 279
    Per-protocol analysis set: Hispanic or Latino | 1 | 1 | 0 | 2
    Per-protocol analysis set: Not Hispanic or Latino | 95 | 89 | 93 | 277
    Per-protocol analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per-protocol set - all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  Participants
    Full analysis set: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Full analysis set: Asian | 7 | 6 | 4 | 17
    Full analysis set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Full analysis set: Black or African American | 10 | 13 | 9 | 32
    Full analysis set: White | 97 | 96 | 103 | 296
    Full analysis set: More than one race | 0 | 0 | 0 | 0
    Full analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0
    Per-protocol analysis set: number analyzed (Participants) | 96 | 90 | 93 | 279
    Per-protocol analysis set: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Per-protocol analysis set: Asian | 7 | 5 | 4 | 16
    Per-protocol analysis set: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Per-protocol analysis set: Black or African American | 8 | 6 | 7 | 21
    Per-protocol analysis set: White | 81 | 79 | 82 | 242
    Per-protocol analysis set: More than one race | 0 | 0 | 0 | 0
    Per-protocol analysis set: Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 4 | 6
  Sweden | 7 | 13 | 10 | 30
  Netherlands | 25 | 19 | 21 | 65
  Singapore | 4 | 2 | 2 | 8
  United States | 52 | 50 | 51 | 153
  Denmark | 0 | 1 | 0 | 1
  United Kingdom | 22 | 28 | 27 | 77
  Germany | 3 | 1 | 1 | 5
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Population: Per-protocol set - all participants who complied with the protocol sufficiently to allow adequate estimation of the treatment effect (including availability of primary pharmacodynamic endpoint assessment and absence of protocol deviations that impact on the treatment effect).
  kilograms per square meter (kg/m^2)
    Full analysis set | 29 (5) | 29 (6) | 31 (5) | 30 (5)
    Per-protocol analysis set: number analyzed (Participants) | 96 | 90 | 93 | 279
    Per-protocol analysis set | 29 (5) | 29 (5) | 30 (5) | 29 (5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pharmacodynamic Response as Assessed by the Inhibition of Platelet Aggregation
Description: The pharmacodynamic response was determined by measuring the inhibition of platelet aggregation, using VerifyNow®. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU). The target of 100 PRU corresponds to 80% inhibition of ADP-induced platelet aggregation. A participant with a PRU of less than 100 starting from 30 minutes after the administration of study treatment and lasting for at least 3 hours was considered a "responder".
Time Frame: From 15 minutes after administration of the subcutaneous injection up to 24 hours
Population: Full Analysis Set - all participants that were randomized and who had study treatment administered.
Measure: Number; unit: Count of participants (i.e., responders)
Groups:
- Selatogrel 8 mg: Selatogrel 8 mg was administered as a single subcutaneous dose.
- Selatogrel 16 mg: Selatogrel 16 mg was administered as a single subcutaneous dose.
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Number analyzed (Participants) | 114 | 115 | 116
Count of participants (i.e., responders) | 102 | 103 | 18
Statistical Analysis 1: Comparison: Selatogrel 8 mg vs Placebo; The study aimed at assessing the efficacy of each selatogrel dose versus placebo. The proportion of responders for each of the two doses of selatogrel was compared to placebo. No imputation was considered for handling missing values; Test type: Superiority; p < 0.0001, Chi-squared — A p-value significance level was set to 0.025, based on an overall Type-I error rate of 0.05 adjusted for multiple comparisons using a Bonferroni approach (two comparisons); Odds Ratio (OR) = 58.9, 97.5% CI 2-sided [22.4 to 154.8]
Statistical Analysis 2: Comparison: Selatogrel 16 mg vs Placebo; The study aimed at assessing the efficacy of each selatogrel dose versus placebo. The proportion of responders for each of the two doses of selatogrel was compared to placebo. No imputation was considered for handling missing values in the main analysis; Test type: Superiority; p < 0.0001, Chi-squared — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 61.2, 97.5% CI 2-sided [23.1 to 162.3]

2. Secondary Outcome: Maximum Selatogrel Plasma Concentration (Cmax)
Description: The Cmax is the peak concentration of selatogrel in the plasma after subcutaneous injection.
  The pharmacokinetic parameters of selatogrel (ACT-246475) were derived by non-compartmental analyses of the plasma concentration-time profiles.
Time Frame: Pre-dose, and from 15 minutes after administration of the subcutaneous injection up to 24 hours
Population: Pharmacokinetic analysis set - all participants that had a selatogrel concentration measurement after administration of study treatment.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 111 | 115
ng/mL | 298 [146 to 868] | 484 [161 to 1030]

3. Secondary Outcome: Time to Reach Maximum Selatogrel Plasma Concentration (Tmax)
Description: Time after subcutaneous injection to reach the maximum observed selatogrel plasma concentration (Cmax).
Time Frame: Pre-dose, and from 15 minutes after administration of the subcutaneous injection up to 24 hours
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 111 | 115
hour | 0.52 [0.38 to 1.05] | 0.53 [0.23 to 2.02]

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve of Selatogrel From Time Zero to 24 Hour Time Point (AUC0-24)
Description: The area under the plasma concentration-time curve is the integral of the concentration-time curve after subcutaneous injection of selatogrel.
  The plasma pharmacokinetic parameters of selatogrel (ACT-246475) were derived by non-compartmental analyses of the plasma concentration-time profiles.
Time Frame: Pre-dose, and from 15 minutes after administration of the subcutaneous injection up to 24 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: hours*ng/mL
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg
Number analyzed (Participants) | 111 | 115
hours*ng/mL | 716 [347 to 1425] | 1358 [487 to 2758]

5. Other Pre Specified Outcome: Number of Participants With a Pharmacodynamic Response as Assessed by the Inhibition of Platelet Aggregation by Site of Treatment Administration (Thigh or Abdomen)
Description: The inhibition of platelet aggregation based on the route of administration, i.e. whether the pharmacodynamic response was different if selatogrel was administered subcutaneously in the thigh or in the abdomen, was analyzed.
  The pharmacodynamic response was determined by measuring the inhibition of platelet aggregation, using VerifyNow®. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU). The target of 100 PRU corresponds to 80% inhibition of ADP-induced platelet aggregation. A participant with a PRU of less than 100 starting from 30 minutes after the administration of study treatment and lasting for at least 3 hours was considered a "responder".
Time Frame: From 15 minutes after administration of the subcutaneous injection up to 24 hours
Population: Full Analysis Set - all participants that were randomized and who had study treatment administered.
Measure: Number; unit: Count of participants (i.e., responders)
Groups:
- Selatogrel 8 mg (Thigh); Selatogrel 8 mg (Abdomen): Selatogrel 8 mg was administered as a single subcutaneous dose.
- Selatogrel 16 mg (Thigh); Selatogrel 16 mg (Abdomen): Selatogrel 16 mg was administered as a single subcutaneous dose.
- Placebo (Thigh); Placebo (Abdomen): Matching placebo was administered as a single subcutaneous dose.
Arm/Group | Selatogrel 8 mg (Thigh) | Selatogrel 8 mg (Abdomen) | Selatogrel 16 mg (Thigh) | Selatogrel 16 mg (Abdomen) | Placebo (Thigh) | Placebo (Abdomen)
Number analyzed (Participants) | 57 | 57 | 57 | 58 | 58 | 58
Count of participants (i.e., responders) | 52 | 50 | 52 | 51 | 11 | 7
Statistical Analysis 1: Comparison: Selatogrel 8 mg (Thigh) vs Selatogrel 8 mg (Abdomen) vs Selatogrel 16 mg (Thigh) vs Selatogrel 16 mg (Abdomen); Test type: Other — Logistic regression (Type III analysis); p = 0.1915, Chi-squared

6. Other Pre Specified Outcome: Number of Participants With a Pharmacodynamic Response as Assessed by the Inhibition of Platelet Aggregation - Sensitivity Analysis
Description: To assess the robustness of results for the pharmacodynamic response, the main analysis was repeated for the per protocol participants. The pharmacodynamic response was determined by measuring the inhibition of platelet aggregation, using VerifyNow®. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU). The target of 100 PRU corresponds to 80% inhibition of ADP-induced platelet aggregation. A participant with a PRU of less than 100 starting from 30 minutes after the administration of study treatment and lasting for at least 3 hours was considered a "responder".
Time Frame: From 15 minutes after administration of the subcutaneous injection up to 24 hours
Population: Per-protocol set
Measure: Number; unit: Count of participants (i.e., responders)
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Number analyzed (Participants) | 96 | 90 | 93
Count of participants (i.e., responders) | 92 | 90 | 16

7. Other Pre Specified Outcome: Change From Baseline in Maximum Platelet Aggregation (MPA) as Measured by Light Transmission Aggregometry (LTA)
Description: Light transmission aggregometry was used as complementary method to the VerifyNow® to evaluate the effect of selatogrel on platelet aggregation. Platelet aggregation was triggered by addition of Adenosine diphosphate (ADP) 20 µM (micromole per liter) and monitored over 6 minutes. Maximum Platelet Aggregation (MPA) to 20 μM ADP was assessed by light transmission aggregometry (LTA), an assay that measures platelet aggregation by determining the amount of light transmitted through a cuvette containing platelet-rich plasma stimulated with 20 µM ADP, relative to platelet-poor plasma (100% light transmittance). A lower MPA % reflects stronger platelet inhibition, whereas a higher MPA % reflects weaker inhibition.
Time Frame: Pre-dose, and from 30 minutes after administration of the subcutaneous injection up to 8 hours
Population: Full Analysis Set - all participants that were randomized and who had study treatment administered.
Measure: Mean (Standard Deviation); unit: percent maximum platelet aggregation (%)
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Number analyzed (Participants) | 114 | 115 | 116
percent maximum platelet aggregation (%)
  Pre-dose: number analyzed (Participants) | 113 | 112 | 115
  Pre-dose | 61.9 (29.79) | 62.4 (31.5) | 65.6 (29.6)
  30 minutes post-dose: number analyzed (Participants) | 114 | 109 | 109
  30 minutes post-dose | 13.1 (12.1) | 13.5 (11.9) | 65.3 (28.0)
  1 hour post-dose: number analyzed (Participants) | 113 | 109 | 114
  1 hour post-dose | 14.5 (14.1) | 15.8 (15.7) | 65.6 (28.0)
  2 hours post-dose: number analyzed (Participants) | 113 | 113 | 114
  2 hours post-dose | 17.0 (12.8) | 16.5 (14.5) | 63.0 (26.8)
  8 hours post-dose: number analyzed (Participants) | 114 | 113 | 112
  8 hours post-dose | 35.4 (25.5) | 32.1 (25.1) | 63.7 (27.0)
Statistical Analysis 1: Comparison: Selatogrel 8 mg vs Placebo; Longitudinal analysis of the treatment effect, from start of treatment to 8 hours after injection; Test type: Other; p < .0001, Mixed Models Analysis; P-value significance level is set to 0.025, i.e. type I error (0.05) adjusted for multiplicity (2 comparisons) using a Bonferroni approach; LS Mean difference with placebo = -27.49, 95% CI 2-sided [-35.4 to -19.6]
Statistical Analysis 2: Comparison: Selatogrel 16 mg vs Placebo; Longitudinal analysis of the treatment effect, from start of treatment up to 8 hours after injection; Test type: Other; p < .0001, Mixed Models Analysis; [statistical method as in outcome 7, analysis 1]; LS Mean difference with placebo = -31.06, 95% CI 2-sided [-39.0 to -23.1]

8. Other Pre Specified Outcome: Number of Participants With Bleeding Events
Description: Treatment-emergent adverse events in the category "Haemorrhage (excluding laboratory terms)" were of special interest and their incidence listed below.
  The role of the Independent Safety Event Committee was to monitor unblinded safety data obtained in the study, with a specific focus on study-drug-related clinically relevant major bleeding events, occurring within 48 hours after dosing (i.e. the treatment period).
Time Frame: From study treatment administration on Day 1 up to 48 hours
Population: The safety analysis set (SAF) included all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Number analyzed (Participants) | 114 | 115 | 116
Participants
  All participants with at least one "bleeding event" | 11 | 5 | 8
  Participants with Trombolysis In Myocardial Infarction (TIMI) major events | 0 | 0 | 0
  Participants with "Bleeding event of moderate intensity" | 0 | 0 | 1
  Participants with "Bleeding event of mild intensity" | 11 | 5 | 7
  Injection site bruising | 3 | 2 | 0
  Contusion | 1 | 1 | 3
  Ecchymosis | 0 | 1 | 0
  Eye contusion | 0 | 1 | 0
  Medical device site bruise | 1 | 0 | 0
  Mouth haemorrhage | 0 | 1 | 0
  Vessel puncture site bruise | 4 | 0 | 3
  Epistaxis | 1 | 0 | 0
  Vessel puncture site haematoma | 1 | 0 | 0
  Petechiae | 0 | 0 | 1
  Vaginal haemorrhage | 0 | 0 | 1
  Wound haemorrhage | 0 | 0 | 1

9. Post Hoc Outcome: Assessments of the Inhibition of Platelet Reactivity at Predefined Time Points
Description: The inhibition of platelet aggregation was determined using VerifyNow®. The VerifyNow® is a point-of-care test measuring platelet reactivity. The results are expressed as P2Y12 reaction units (PRU). After single-dose administration the inhibition of platelet aggregation was measured at pre-defined timepoints to observe the platelet reactivity and aggregation over a 24-hour timeperiod. A lower PRU reflects lower platelet reactivity, whereas a higher PRU reflects higher platelet reactivity.
Time Frame: Pre-dose (baseline) up to 24 hours post-dose injection
Population: Full Analysis Set - all participants that were randomized and who had study treatment administered.
Measure: Mean (95% Confidence Interval); unit: P2Y12 reaction units
Arm/Group | Selatogrel 8 mg | Selatogrel 16 mg | Placebo
Number analyzed (Participants) | 114 | 115 | 116
P2Y12 reaction units
  Baseline (pre-dose) | 156.1 [142.9 to 169.3] | 156.2 [142 to 170.5] | 155.2 [141.9 to 168.6]
  15 minutes post-dose: number analyzed (Participants) | 111 | 110 | 108
  15 minutes post-dose | 10.1 [5.3 to 14.9] | 4.5 [2.6 to 6.4] | 163.3 [149.5 to 177.2]
  30 minutes post-dose: number analyzed (Participants) | 110 | 110 | 108
  30 minutes post-dose | 7.9 [3.6 to 12.2] | 5.3 [3.4 to 7.2] | 162.2 [147.9 to 176.4]
  1 hour post-dose: number analyzed (Participants) | 108 | 107 | 113
  1 hour post-dose | 9.7 [4.5 to 14.8] | 3.5 [2.6 to 4.5] | 161.8 [148.6 to 175.0]
  2 hours post-dose: number analyzed (Participants) | 110 | 107 | 113
  2 hours post-dose | 12.4 [7.0 to 17.8] | 5.7 [3.7 to 7.6] | 162.0 [148.5 to 175.4]
  4 hours post-dose: number analyzed (Participants) | 109 | 109 | 112
  4 hours post-dose | 30.1 [22.9 to 37.3] | 11.4 [7.8 to 14.9] | 162.4 [148.8 to 176.0]
  8 hours post-dose: number analyzed (Participants) | 110 | 107 | 111
  8 hours post-dose | 88.1 [76.6 to 99.7] | 47.3 [38.9 to 55.6] | 164.1 [150.6 to 177.6]
  24 hours post-dose: number analyzed (Participants) | 111 | 111 | 112
  24 hours post-dose | 144.2 [130.2 to 158.1] | 128.6 [116.3 to 140.9] | 153.3 [139.4 to 167.2]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded up to 35 days after the single subcutaneous selatogrel dose administration. Treatment period: Treatment emergent adverse events were those adverse events with onset and up to 48 hours after study treatment administration. The follow-up period started on Day 3 and ended with the safety follow-up telephone call 35 days after selatogrel administration. During the follow-up period the participants continued to be observed. No interventions were performed.
Groups:
- Treatment Period - Selatogrel 8 mg: In the treatment period 8 mg of selatogrel was administered via a single subcutaneous injection either in the abdomen or the thigh.
- Treatment Period - Selatogrel 16 mg: In the treatment period 16 mg of selatogrel was administered via a single subcutaneous injection either in the abdomen or the thigh.
- Treatment Period - Placebo: In the treatment period placebo matching selatogrel was administered via a single subcutaneous injection either in the abdomen or the thigh.
- Follow-up Period - Selatogrel 8 mg: Participants that had been administered a single subcutaneous injection containing 8 mg selatogrel in the treatment period were followed-up for adverse events after the treatment period. The follow-up period started on Day 3 and ended with a telephone call or visit on Day 35.
- Follow-up Period - Selatogrel 16 mg: Participants that had been administered a single subcutaneous injection containing 16 mg selatogrel were followed-up for adverse events after the treatment period. The follow-up period started on Day 3 and ended with a telephone call or visit on Day 35.
- Follow-up Period - Placebo: Participants that had been administered a single subcutaneous injection containing placebo matching selatogrel were followed-up for adverse events after the treatment period. The follow-up period started on Day 3 and ended with a telephone call or visit on Day 35.
Arm/Group | Treatment Period - Selatogrel 8 mg | Treatment Period - Selatogrel 16 mg | Treatment Period - Placebo | Follow-up Period - Selatogrel 8 mg | Follow-up Period - Selatogrel 16 mg | Follow-up Period - Placebo
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/115 | 0/116 | 1/114 | 0/115 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/115 | 0/116 | 5/114 | 1/115 | 1/116
Other Adverse Events (participants affected / at risk) | 36/114 | 26/115 | 25/116 | 13/114 | 10/115 | 13/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period - Selatogrel 8 mg (N=114) | Treatment Period - Selatogrel 16 mg (N=115) | Treatment Period - Placebo (N=116) | Follow-up Period - Selatogrel 8 mg (N=114) | Follow-up Period - Selatogrel 16 mg (N=115) | Follow-up Period - Placebo (N=116)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant was hospitalized 26 days after study treatment administration.
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Participant was hospitalized 12 days after study treatment administration.
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant was hospitalized 30 days after study treatment administration.
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant was hospitalized 12 days after study treatment administration.
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant was hospitalized 14 days after study treatment administration.
Myocardial infarctions (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Participant was hospitalized 18 days after study treatment administration.
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant died 18 days after study treatment administration.
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant died 18 days after study treatment administration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period - Selatogrel 8 mg (N=114) | Treatment Period - Selatogrel 16 mg (N=115) | Treatment Period - Placebo (N=116) | Follow-up Period - Selatogrel 8 mg (N=114) | Follow-up Period - Selatogrel 16 mg (N=115) | Follow-up Period - Placebo (N=116)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruise (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 4 (6) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site erythema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ECG P wave inverted (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 10 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Blood was collected with phenylalanine-proline-arginine-chloromethyl ketone as anticoagulant. Any direct comparison of absolute PRU values obtained in this study with those published from studies of other P2Y12 inhibitors should take this into account.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03384966/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT03384966/SAP_001.pdf